CLINICAL TRIAL: NCT06680258
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study of TPST-1120 in Combination With Atezolizumab Plus Bevacizumab Compared With Placebo Plus Atezolizumab Plus Bevacizumab in Patients With Unresectable or Metastatic Hepatocellular Carcinoma (HCC) Not Previously Treated With Systemic Therapy
Brief Title: A Study of TPST-1120 With Atezolizumab Plus Bevacizumab in Patients With Unresectable or Metastatic HCC Not Previously Treated With Systemic Therapy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tempest Therapeutics (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPST-1120-301
Record Dates: First submitted 2024-11-04; First posted 2024-11-08 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Hepatocellular carcinoma; liver cancer; metastatic; atezolizumab; bevacizumab; advanced; unresectable; PD-L1; b-catenin; CTNNB1
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Neoplasm Metastasis | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Arm (Experimental): TPST-1120 600 mg by mouth (PO) twice daily (BID) with atezolizumab 1200 mg intravenously (IV) every 3 weeks (Q3W) and bevacizumab 15 mg/kg IV Q3W
  Interventions: Drug: TPST-1120; Biological: Atezolizumab; Biological: Bevacizumab
- Control Arm (Active Comparator): Placebo tablets PO BID with atezolizumab 1200 mg IV Q3W and bevacizumab 15 mg/kg IV Q3W
  Interventions: Biological: Atezolizumab; Biological: Bevacizumab

INTERVENTIONS:
Drug: TPST-1120 — TPST-1120 is an orally administered competitive antagonist of peroxisome proliferator-activated receptor α (PPARα)
  Arms: Active Arm
Biological: Atezolizumab — Atezolizumab is an IV administered biologic.
Biological: Bevacizumab — Bevacizumab is an IV administered biologic.

SUMMARY:
The goal of this clinical trial is to determine if TPST-1120 in combination with atezolizumab and bevacizumab helps patients to live longer compared to atezolizumab and bevacizumab alone (the standard of care treatment) in adult patients with hepatocellular carcinoma that cannot be removed by surgery or has spread outside of the liver (called metastatic). The trial also will study the safety and side effects of the drug combination compared to the standard of care treatment. Other questions the trial aims to answer include:

1. Does TPST-1120 in combination with atezolizumab and bevacizumab improve the time that patients are alive and cancer is not growing (progression free survival) compared to atezolizumab and bevacizumab
2. Does TPST-1120 in combination with atezolizumab and bevacizumab improve the shrinking of cancer (the overall response rate) compared to atezolizumab and bevacizumab

Trial participants will be randomly assigned to take one of the following:

1. TPST-1120 3 tablets (600 mg) by mouth twice a day every day along with atezolizumab 1200 mg intravenously every 3 weeks and bevacizumab 15 mg/kg intravenously every 3 weeks
2. Placebo (look-alike that does not contain study drug) 3 tablets by mouth twice a day every day along with atezolizumab 1200 mg intravenously once every 3 weeks and bevacizumab 15 mg/kg intravenously once every 3 weeks

Trial participants will receive routine and trial-specific cancer care from their study doctor including

* visits to the clinic every 3 weeks for physical examination, labs and questions about health and symptoms
* measurement of their cancer by CT scan every 9 weeks.

Trial participants can stop study treatment at any time they choose and for any reason. They also can continue to receive study treatment for as long as the treatment is controlling cancer growth and they are tolerating the drug effects.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, multicenter, double-blind, Pbo-controlled study of TPST-AB versus Pbo-AB in patients with unresectable or metastatic HCC not previously treated with systemic therapy.

The study will consist of a screening period, a treatment period, and a follow-up period.

The purpose of this study is to measure the safety and efficacy of TPST-1120 in combination with atezolizumab plus bevacizumab compared with placebo plus atezolizumab plus bevacizumab in patients with unresectable or metastatic HCC who have received no prior systemic treatment. Study details include:

* Study duration: until death, loss to follow-up, withdrawal of consent, or study termination, whichever occurs first]
* Treatment duration: until unacceptable toxicity or loss of clinical benefit
* Visit frequency: every 21 days

Approximately 740 patients are planned to be randomized and enrolled.

Eligible patients will be randomized in a 1:1 ratio to receive study intervention with the combination of TPST-AB or Pbo-AB as follows:

* Active arm: TPST-1120 600 mg per os (PO) twice daily (BID) with atezolizumab 1200 mg intravenously (IV) every 3 weeks (Q3W) and bevacizumab 15 mg/kg IV Q3W
* Control arm: Placebo PO BID with atezolizumab 1200 mg IV Q3W and bevacizumab 15 mg/kg IV Q3W

Patients may continue to receive study intervention until unacceptable toxicity or loss of clinical benefit as determined by the investigator after an integrated assessment of radiographic and biochemical data, and clinical status (e.g., symptomatic deterioration such as pain secondary to disease). In the absence of unacceptable toxicity, patients who meet criteria for disease progression per RECIST v1.1 while receiving study intervention will be permitted to continue the study intervention if they meet all of the following criteria:

* Evidence of clinical benefit, as determined by the investigator following a review of all available data
* Absence of symptoms and signs (including laboratory values, such as new or worsening hypercalcemia) indicating unequivocal progression of disease
* Absence of decline in Eastern Cooperative Oncology Group (ECOG) performance status that can be attributed to disease progression
* Absence of tumor progression at critical anatomical sites (e.g., leptomeningeal disease) that would require urgent alternative medical intervention

Patients will undergo tumor assessments at baseline and then, timed from initiation of treatment, every 9 weeks (± 1 week) for the first 54 weeks and then every 12 weeks (± 2 weeks) thereafter, regardless of study treatment holds or delays.

Patients who discontinue study intervention will return to the clinic for an End-of-Treatment (EOT) visit no more than 30 days after the final dose of study intervention and prior to the initiation of any new anti-cancer therapy/regimen.

After treatment discontinuation, information on survival follow-up and any new anti-cancer therapies started will be collected approximately every 3 months until death, withdrawal of consent or study completion.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age ≥ 18 years at the time of signing ICF
3. HCC diagnosis confirmed by histology/cytology or clinically by the American Association for the Study of Liver Diseases (AASLD) criteria in cirrhotic patients

   a) Patients without cirrhosis require histological confirmation of diagnosis.
4. Unresectable or metastatic disease not amenable to curative intent surgical and/or locoregional therapies

   a) Patients who have progressed after surgical and/or locoregional therapy for HCC are eligible.
5. No prior systemic therapy (including systemic investigational agents) for HCC
6. At least one measurable (per RECIST v1.1) untreated lesion

   1. Patients who received prior local therapy (e.g., radiofrequency ablation, percutaneous ethanol or acetic acid injection, cryoablation, high-intensity focused ultrasound, transarterial chemoembolization, transarterial embolization, etc.) are eligible provided the target lesion(s) have not been previously treated with local therapy or the target lesion(s) within the field of local therapy have subsequently progressed in accordance with RECIST v1.1.
7. Resolution of any acute, clinically significant treatment-related toxicity from prior therapy to Grade ≤ 1 prior to study entry, except for alopecia
8. ECOG performance status of 0 or 1within 7 days prior to randomization
9. Child-Pugh class A within 7 days prior to randomization
10. Adequate organ and bone marrow function, as defined in protocol (obtained within 7 days prior to randomization unless otherwise specified)
11. Negative human immunodeficiency virus (HIV) test at screening
12. Documented virology status of hepatitis, as confirmed by screening tests for HBV and HCV a) For patients with active HBV: HBV DNA < 500 IU/mL during screening, initiation of anti-HBV treatment at least 14 days prior to randomization and willingness to continue anti-HBV treatment during the study (per local standard of care; e.g., nucleos(t)ide analogues)
13. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use 2 methods of effective contraception, including at least one method with a failure rate of < 1% per year, during the treatment period and for at least 5 months after the last dose of atezolizumab, 6 months after the last dose of bevacizumab, or 3 months after the last dose of TPST-1120/Pbo, whichever is latest. Women must refrain from donating eggs during this same period.
14. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm during the treatment period and for 6 months after the final dose of bevacizumab or 3 months after the last dose of TPST-1120/Pbo, whichever is latest.
15. Consent to submit and provide mandatory tumor sample for central determination of PD L1 status. This may be an archived tumor sample (taken ≤ 3 years) or a fresh tumor biopsy if archived tissue is not available. Tissue specimens must be of sufficient quantity and quality for defining tumor PD-L1.

Exclusion Criteria

1. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
2. History of malignancy other than HCC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, low grade prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer
3. Patients with symptomatic, untreated, or actively progressing central nervous system (CNS) metastases, or any history of leptomeningeal cancer, are not eligible.
4. Metastatic disease that involves major airways or blood vessels, or centrally located mediastinal tumor masses (< 30 mm from the carina)

   a) Patients with vascular invasion of the portal or hepatic veins may be enrolled.
5. Untreated or incompletely treated esophageal and/or gastric varices

   1. Patients must undergo an esophagogastroduodenoscopy (EGD), and all size of varices (small to large) must be treated with definitive therapy (e.g., banding) per local standard of care prior to study enrollment.
   2. Screening EGD does not need to be performed if EGD and definitive variceal treatment were previously completed no more than 6 months prior to initiation of study intervention.
6. Grade ≥ 3 hemorrhage or bleeding event within 8 weeks prior to initiation of study intervention
7. History of hemoptysis (≥ 2.5 mL of bright red blood per episode) within 1 month prior to initiation of study intervention
8. Inadequately controlled hypertension, defined as systolic blood pressure (BP) >150 mmHg and/or diastolic BP > 100 mmHg, based on an average of at least 3 readings at 2 or more sessions

   a) Anti-hypertensive therapy to achieve these parameters is allowed.
9. Prior history of hypertensive crisis or hypertensive encephalopathy
10. History of hepatic encephalopathy
11. History of abdominal or tracheoesophageal fistula, gastrointestinal (GI) perforation, or intra-abdominal abscess within 6 months prior to initiation of study intervention
12. History of intestinal obstruction and/or symptoms of GI obstruction, including subocclusive or occlusive syndrome related to the underlying disease, or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding prior to initiation of study intervention
13. Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture
14. History of a clinically significant intra-abdominal inflammatory process within 6 months prior to initiation of study intervention, including, but not limited to, peptic ulcer disease, diverticulitis, or colitis
15. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (≥ once monthly)
16. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to initiation of study intervention; or abdominal surgery, abdominal interventions or significant abdominal traumatic injury within 60 days prior to initiation of study intervention; or anticipation of need for major surgical procedure during the course of the study or non-recovery from side effects of any such procedure
17. Known active tuberculosis (TB)
18. Uncontrolled tumor-related pain
19. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

    a) Patients with a history of controlled hypothyroidism or controlled Type 1 diabetes are eligible if on stable treatment.
20. Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study intervention, unstable arrhythmia, or unstable angina
21. Severe infection within 4 weeks prior to initiation of study intervention, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that, in the opinion of the investigator, could impact patient safety
22. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
23. QTc interval (calculated using Fridericia method) > 470 ms
24. Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
25. Treatment with locoregional therapy to liver is not allowed within 28 days prior to initiation of study treatment, including radiofrequency ablation, percutaneous ethanol or acetic acid injection, cryoablation, high-intensity focused ultrasound, transarterial chemoembolization, transarterial yttrium-90 embolization, transarterial bland embolization (note that locoregional liver treatment prior to 28 days is allowed)
26. External beam radiation therapy is not allowed within 28 days prior to initiation of study treatment with exception of (i) whole abdominal or pelvic radiotherapy are not allowed within 60 days, (ii) palliative radiotherapy to bone is not allowed within 7 days, and (iii) stereotactic radiotherapy to CNS lesions is not allowed within 7 days of initiation of study treatment.

    a) Washout of transarterial Y90 embolization to liver is 28 days as per exclusion criterion #33
27. Treatment with fibrates (e.g., gemfibrozil, fenofibrate) within 28 days prior to initiation of study intervention
28. Use of strong CYP3A4 inhibitors (e.g., atazanavir, clarithromycin, grapefruit juice, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, and voriconazole) or strong CYP3A4 inducers (e.g., barbiturates, efavirenz, nevirapine, ritonavir, and topiramate) within 7 days of initiation of study intervention (30 days for enzalutamide and apalutamide)
29. Current or recent (≤ 10 days prior to initiation of study intervention) use of a) Aspirin (≥ 325 mg/day) or treatment with clopidogrel, dipyridamole, ticlopidine, or cilostazol b) Full dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic (as opposed to prophylactic) purpose i) Prophylactic anticoagulation for the patency of venous access devices is allowed, provided the activity of the agent results in an INR < 1.5 × ULN and aPTT is within normal limits within 14 days prior to initiation of study intervention.

ii) For prophylactic use of anticoagulants or thrombolytic therapies, the approved dose per local label may be used.

31. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin (IL)-2) within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to initiation of study intervention 32. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids > 10 mg daily prednisone equivalent, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor (TNF)-α agents) within 2 weeks prior to initiation of study intervention, or anticipation of need for systemic immunosuppressive medication during study intervention, with the following exceptions:

1. Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Medical Monitor confirmation has been obtained.
2. Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for COPD or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal Prior/Concurrent Clinical Study Experience 33. Inability to receive study intervention orally in intact form or any condition that may prevent adequate absorption of oral study intervention including refractory nausea and vomiting, uncontrolled diarrhea, malabsorption, significant small bowel resection or gastric bypass surgery, or use of feeding tubes 34. Female patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | The time from randomization to death from any cause up to 60 months.
  Overall survival (OS), defined as the time from randomization to death from any cause up to 60 months.

SECONDARY OUTCOMES:
Progression free survival | The time from randomization to first occurence of disease progression or death from any cause (whichever occurs first) up to 60 months.
  Defined as the time from randomization to the first occurrence of disease progression or death from any cause (whichever occurs first) up to 60 months, as determined by investigator-assessment, per the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1

IPD SHARING:
Plan to Share IPD: No